CLINICAL TRIAL: NCT03243630
Title: Effects of Flavors on Nicotine Reinforcement in Smokers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2000021591; 1P50DA036151-01 (NIH)
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Results first posted 2020-11-13 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Menthol

STUDY DESIGN:
Intervention Model Description: Mixed-effects models will be used to test the study hypotheses. These models allow for different numbers of observations per subject, use all available data on each subject, and are unaffected by randomly missing data.
Who Masked: Participant, Investigator
Masking Description: The participant and medical professional will be blinded to the condition per day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Menthol e-liquid (Placebo Comparator): Menthol Flavor + IV saline Menthol Flavor + IV nicotine (0.25mg/70kg) Menthol Flavor + IV nicotine (0.5mg/70kg)
  Interventions: Drug: IV nicotine; Drug: Menthol flavor; Drug: green apple; Drug: green apple and menthol
- green apple e-liquid (Active Comparator): Green apple + IV saline Green apple + IV nicotine (0.25mg/70kg) Green apple + IV nicotine (0.5mg/70kg)
  Interventions: Drug: IV nicotine; Drug: Menthol flavor; Drug: green apple; Drug: green apple and menthol
- green apple and menthol e-liquid (Active Comparator): Green apple and menthol + IV saline Green apple and menthol + IV nicotine (0.25mg/70kg) Green apple and menthol + IV nicotine (0.5mg/70kg)
  Interventions: Drug: IV nicotine; Drug: Menthol flavor; Drug: green apple; Drug: green apple and menthol

INTERVENTIONS:
Drug: IV nicotine — Subjects in each arm will receive three infusions in a random order one hour apart. The infusions will be saline, 0.25mg/70kg and 0.5mg/70kg
  Other Names: nicotine, e-liquid
Drug: Menthol flavor — American e-liquids' menthol flavor used in e-cigarettes will be used as the placebo comparator
  Other Names: menthol American e-liquids
Drug: green apple — green apple will be added to the menthol flavor
  Other Names: green apple American e-liquids
Drug: green apple and menthol — menthol and green apple will be the active intervention
  Other Names: green apple and menthol flavor American e-liquids

SUMMARY:
To examine the acute reinforcing effects of menthol, a fruit flavor (green apple) or a fruit flavor plus menthol, alone or in combination with nicotine in smokers. Flavors will be administered by inhalation via electronic cigarettes (e-cigarettes) and nicotine will be administered intravenously. The reinforcing drug effects will be measured with the drug effects questionnaire (DEQ).

DETAILED DESCRIPTION:
This is a proposed double-blind, crossover study that enrolls young adult smokers who prefer menthol cigarettes. The study will consist of an adaptation session and three test sessions. In the adaptation session, participants will practice using the e-cigarette by sampling the flavors to be used in the test sessions. The test sessions will be performed following overnight abstinence from tobacco. Across the three test sessions, participants will be assigned to a random sequence of the three different e-cigarette conditions: menthol, green apple or menthol plus green apple, a different flavor condition for each test session. In each test session, just after the assigned flavor is delivered via the e-cigarette, participants will receive a random order of one intravenous delivery of saline, and two intravenous deliveries of nicotine (3.6 mcg/kg and 7 mcg/kg or 0.25 mg/70 kg and 0.5 mg/70kg), one hour apart. The test sessions will be performed at least 24 hours apart to minimize carryover nicotine effects. The main outcome measure will be subjective drug effects as measured with the Drug Effects Questionnaire (DEQ). Other outcomes include cardiovascular measures, cognitive performance, and self-report measures of nicotine withdrawal and craving. Cardiovascular measures include heart rate, systolic and diastolic blood pressure. Cognitive performance will be assessed with the Stroop test, mathematical processing test (MPT), and continuous performance test (CPT). Nicotine withdrawal measures will be measured with the Minnesota Nicotine Withdrawal Symptom Checklist (M-NWSC) and the Brief Questionnaire on Smoking Urges (BQSU).

ELIGIBILITY:
Inclusion Criteria:

Female and male mentholated cigarette smokers, aged 18 to 30 years; history of smoking for the past 12 months, at least one cigarette per day; smoking status is verified with urinary cotinine levels above 10 ng/ml; not seeking treatment for nicotine dependence at the time of study entry in good health as verified by medical history, screening examination, and screening laboratory tests; for women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

History of major medical illnesses that the physician investigator deems as contraindicated for the patient to be in the study; regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics); psychiatric diagnosis and / or treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia or panic disorder in the past month; abuse of alcohol or any other recreational or prescription drugs in the past 30 days; any allergy to propylene glycol or menthol; and 6) aversion to green apple flavor.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D.Ph.D., Principal Investigator — Yale University
Locations (1):
- Veterans Affairs, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 26 subjects were eligible for participation with 24 randomized after completion of the adaptation session. Reasons for exclusion after adaptation session included poor venous access (n=1) and a positive drug screen (n=1).
Pre-assignment Details: A total of 26 subjects were eligible for participation with 24 randomized after completion of the adaptation session.
Groups:
- Study Cohort: In each test session, the flavor was randomly assigned and delivered via the e-cigarette. Then, participants were randomly assigned to receive one intravenous delivery of saline, and two intravenous deliveries of nicotine (3.6 mcg/kg and 7 mcg/kg or 0.25 mg/70 kg and 0.5 mg/70kg), one hour apart.
  Menthol Flavor + IV saline Menthol Flavor + IV nicotine (0.25mg/70kg) Menthol Flavor + IV nicotine (0.5mg/70kg)
  Green Apple Flavor + IV saline Green Apple Flavor + IV nicotine (0.25mg/70kg) Green Apple Flavor + IV nicotine (0.5mg/70kg)
  Menthol plus Green Apple Flavor + IV saline Menthol plus Green Apple Flavor + IV nicotine (0.25mg/70kg) Menthol plus Green Apple Flavor + IV nicotine (0.5mg/70kg)
Period: Overall Study
Arm/Group | Study Cohort
Started | 24
Menthol E-liquid Saline | 22
Menthol E-liquid Higher | 22
Menthol E-liquid Lower | 22
Green Apple E-liquid Saline | 20
Green Apple E-liquid Higher | 20
Green Apple E-liquid Lower | 20
Green Apple and Menthol E-liquid Saline | 21
Green Apple and Menthol E-liquid Higher | 21
Green Apple and Menthol E-liquid Lower | 21
Completed | 22
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: The baseline characteristics has been provided for the entire study. Test sessions were randomized by arm, each test session was a different arm.
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 15
  Caucasian | 7
  Other | 4
  Hispanic ethnicity | 6
Fagerstrom Test of Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — The test was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence.
  In scoring the Fagerstrom Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. A score of 3 greater indicates dependence on nicotine The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
  units on a scale | 3.2 (2.1)
Average cigarette consumption per day [Mean (Standard Deviation); unit: cigarette] | 8.3 (4.5)
Years of smoking [Mean (Standard Deviation); unit: years] | 13.2 (2.4)
serum cotinine level [Mean (Standard Deviation); unit: ng/ml] | 194.4 (123.8)
Positive THC at screen [Number; unit: participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: The Reinforcing Drug Effects Will be Measured With the Drug Effects Questionnaire (DEQ).
Description: The (DEQ) Drug Effects Questionnaire has eleven questions with a minimum score of 0 to a maximum score of 100.
  Peak values from each time points were calculated for the change in the intensity of positive subjective effects as measured with these peak values for like and want more were averaged to obtain a summary score to represent the feel "good drug effects" composite factor. Higher scores for each DEQ represent greater endorsement of that subjective effect (e.g., on the "like drug" scale a response of 90 represents greater liking than a response of 50).
Time Frame: up to 3 hours per test session.
Population: Data was analyzed as Intention to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Menthol E-liquid | Green Apple E-liquid | Green Apple and Menthol E-liquid
Number analyzed (Participants) | 22 | 20 | 20
units on a scale
  Higher Nicotine : Max_Cool: number analyzed (Participants) | 22 | 18 | 20
  Higher Nicotine : Max_Cool | 43.18 (26.49) | 26.22 (25.83) | 25.20 (21.38)
  Higher Nicotine : Max_Like: number analyzed (Participants) | 22 | 18 | 20
  Higher Nicotine : Max_Like | 56.00 (28.14) | 53.44 (28.03) | 50.80 (34.69)
  Higher Nicotine : Max_Dislike: number analyzed (Participants) | 22 | 18 | 20
  Higher Nicotine : Max_Dislike | 24.36 (29.86) | 25.88 (31.41) | 20.80 (27.59)
  Higher Nicotine : Max_Craving: number analyzed (Participants) | 22 | 18 | 20
  Higher Nicotine : Max_Craving | 41.27 (35.29) | 46.00 (36.57) | 49.90 (36.90)
  Lower Nicotine: Max_Cool: number analyzed (Participants) | 22 | 19 | 20
  Lower Nicotine: Max_Cool | 33.27 (26.16) | 17.47 (22.45) | 25.90 (26.66)
  Lower Nicotine: Max_Like: number analyzed (Participants) | 22 | 19 | 20
  Lower Nicotine: Max_Like | 46.09 (31.02) | 50.11 (30.44) | 42.90 (32.40)
  Lower Nicotine: Max_Dislike: number analyzed (Participants) | 22 | 19 | 20
  Lower Nicotine: Max_Dislike | 13.63 (17.48) | 13.36 (21.65) | 14.50 (23.45)
  Lower Nicotine: Max_Craving | 48.00 (35.69) | 53.16 (37.34) | 49.00 (37.95)
  Saline: Max_Cool | 31.45 (21.97) | 15.50 (20.56) | 24.60 (22.96)
  Saline: Max_Like | 33.00 (30.67) | 35.80 (31.65) | 32.90 (27.04)
  Saline: Max_Dislike | 8.72 (12.64) | 15.50 (23.75) | 14.40 (23.79)
  Saline: Max_Craving | 46.09 (39.44) | 57.70 (36.60) | 55.80 (38.24)

ADVERSE EVENTS:
Time Frame: The SAFTEE is a technique for the systematic assessment of side effects in clinical trials developed by National Institute of Mental Health This was used before each Test Session and after each test session participants were observed no more than one month. There were no adverse events reported.
Description: The SAFTEE is a technique for the systematic assessment of side effects in clinical trials developed by National Institute of Mental Health
Arm/Group | Menthol E-liquid | Green Apple E-liquid | Green Apple and Menthol E-liquid
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT03243630/Prot_SAP_000.pdf